CLINICAL TRIAL: NCT00413634
Title: A Phase II, Open-label, Multicentre, Pharmacokinetic, Pharmacodynamic and Safety Study of Anagrelide Hydrochloride in Young (18-50 Years) and Elderly (≥ 65 Years) Patients With Essential Thrombocythaemia.
Brief Title: The Pharmacokinetics of Anagrelide in Elderly and Young Patients With Essential Thrombocythaemia (ET)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPD422-203; 2004-004058-20 (EudraCT Number)
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Essential Thrombocythaemia
MeSH Terms: conditions — Thrombocythemia, Essential | interventions — anagrelide

ARMS (2):
- Younger Participants (18-50 years) (Experimental)
  Interventions: Drug: anagrelide hydrochloride
- Elderly Participants (≥65 years) (Experimental)
  Interventions: Drug: anagrelide hydrochloride

INTERVENTIONS:
Drug: anagrelide hydrochloride — Anagrelide hydrochloride 0.5 mg per capsule; participants will be stable on an anagrelide treatment regimen and will take capsules from their own prescription except on the PK day when the participant specific anagrelide dose will be administered from a controlled study specific supply.
  Arms: Younger Participants (18-50 years)
Drug: anagrelide hydrochloride — Anagrelide hydrochloride 0.5 mg per capsule; participants will be stable on an anagrelide regimen and will take capsules from their own prescription except on the PK day when the participant specific anagrelide dose will be administered from a controlled study specific supply.
  Arms: Elderly Participants (≥65 years)

SUMMARY:
Age related differences in response to a drug could arise from variation in pharmacokinetic (PK) and/or pharmacodynamic (PD) profiles between age groups. Whilst the efficacy and safety profile of anagrelide is well established through a well-documented clinical trial programme in patients of all ages, no formal studies have been carried out to investigate whether the PK profile of anagrelide and its metabolites is altered with age.

This study is designed to allow comparisons to be made in terms of pharmacokinetics of anagrelide and its metabolites between elderly (≥ 65 years) and young (18-50 years) ET patients

ELIGIBILITY:
Inclusion Criteria:

* Young patients aged 18-50 years inclusive or Elderly patients aged 65 years and over
* Patients must have a confirmed diagnosis of ET.
* Currently receiving anagrelide hydrochloride at a stable maintenance dose < 5 mg/day for at least 4 weeks.

Exclusion Criteria:

* Diagnosis of any other myeloproliferative disorder.
* Current use of tobacco in any form (e.g. smoking or chewing)
* Treatment with any known enzyme altering agents (barbiturates, phenothiazines, cimetidine etc.) within 30 days prior to or during the study.
* Patients for whom use of another cytoreductive agent in addition to anagrelide is considered necessary for control of platelet count.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-11-13 (Actual); Primary Completion 2008-01-22 (Actual); Study Completion 2008-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- Hospitl Del Mar, Barcelona, Spain
- Sweden (3):
  - Quintiles Hermelinen, Luleå
  - Uppsala Akademiska Sjukhus, Uppsala
  - Quintiles AB Phase I Unit, Uppsala
- Belfast City Hospital, Belfast, United Kingdom

REFERENCES:
- [Derived] Besses C, Zeller W, Alvarez-Larran A, Coll R, Troy S, Purkayastha J, Martin P, Freitag C. Pharmacokinetics and tolerability of anagrelide hydrochloride in young (18 - 50 years) and elderly (>/= 65 years) patients with essential thrombocythemia. Int J Clin Pharmacol Ther. 2012 Nov;50(11):787-96. doi: 10.5414/CP201711. PMID 22943924
- See also: FDA-approved Label — http://www.accessdata.fda.gov/drugsatfda_docs/label/2009/020333s015lbl.pdf
- See also: FDA Recall Information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were between 18-50 years (young) and 65 or older (elderly) with a diagnosis of essential thrombocythemia (ET) and receiving a stable dose of anagrelide <=5mg/day for at least 4 weeks.
Pre-assignment Details: The study comprised four phases: Screening (patients take their normal regimen of anagrelide), a run-in period (patients divided their normal anagrelide daily dose equally into two daily doses), Pharmacokinetics (PK) sampling day (patients take normal morning dose), and follow-up (patients were contacted by phone 30 days after PK visit).
Groups:
- Agrylin (Young): Anagrelide hydrochloride in ages 18-50 years
- Agrylin (Elderly): Anagrelide hydrochloride in ages 65 and older
Period: Overall Study
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Agrylin (Young) | Agrylin (Elderly) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 0 | 12
  >=65 years | 0 | 12 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (8.4) | 69.2 (3.0) | 54.2 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 3 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 5 | 10 | 15
  United Kingdom | 2 | 1 | 3
  Spain | 1 | 1 | 2
  Sweden | 2 | 0 | 2
  Serbia | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Agrylin
Time Frame: over 1 day
Population: PK population (defined as all patients with post-dose drug concentration data)
Measure: Geometric Mean (Standard Deviation); unit: ng/ml
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
ng/ml | 2.66 (0.99) | 3.63 (1.44)
Statistical Analysis 1: Comparison: Agrylin (Young) vs Agrylin (Elderly); Test type: Superiority or Other; p = 0.092, ANOVA

2. Secondary Outcome: Platelet Count
Description: Platelet counts in patients with ET receiving Agrylin
Time Frame: over 1 day
Population: Safety population (defined as all patients who received study treatment)
Measure: Mean (Standard Deviation); unit: x 1,000,000,000/L
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
x 1,000,000,000/L
  Baseline | 488.8 (167.4) | 548.5 (278.7)
  2 hours post-dose | 487.9 (168.1) | 539.2 (258.6)
  12 hours post-dose | 473.2 (146.0) | 540.3 (263.6)

3. Secondary Outcome: Heart Rate
Description: Heart rates in patients with ET receiving Agrylin
Time Frame: over 1 day
Population: Safety population
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
beats/min
  Baseline | 74.0 (9.6) | 70.3 (8.4)
  0.5 hours post-dose | 72.4 (8.9) | 77.7 (13.5)
  1 hour post-dose | 75.8 (5.5) | 80.6 (11.7)
  1.5 hours post-dose | 78.1 (7.7) | 82.7 (12.9)
  2 hours post-dose | 74.3 (7.0) | 81.2 (13.8)
  4 hours post-dose | 75.0 (5.5) | 74.7 (13.7)
  6 hours post-dose | 75.9 (8.6) | 76.9 (11.4)
  8 hours post-dose | 75.5 (6.7) | 76.3 (10.1)
  12 hours post-dose | 73.2 (6.0) | 71.9 (8.1)

4. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of Agrylin
Time Frame: over 1 day
Population: PK population
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
hours | 1.11 (0.39) | 1.14 (0.91)
Statistical Analysis 1: Comparison: Agrylin (Young) vs Agrylin (Elderly); Test type: Superiority or Other; p = 0.857, ANOVA

5. Primary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC) of Agrylin
Time Frame: over 1 day
Population: PK population
Measure: Geometric Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
ng.h/ml | 6.4 (2.4) | 10.3 (4.0)
Statistical Analysis 1: Comparison: Agrylin (Young) vs Agrylin (Elderly); Test type: Superiority or Other; p = 0.013, ANOVA

6. Primary Outcome: Terminal Half-life (T 1/2) of Agrylin
Time Frame: over 1 day
Population: PK population
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
hours | 1.3 (0.4) | 1.4 (0.3)
Statistical Analysis 1: Comparison: Agrylin (Young) vs Agrylin (Elderly); Test type: Superiority or Other; p = 0.378, ANOVA

7. Primary Outcome: Total Clearance (CL/F) of Agrylin
Time Frame: over 1 day
Population: PK population
Measure: Geometric Mean (Standard Deviation); unit: L/h
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
L/h | 156 (73) | 97 (70)
Statistical Analysis 1: Comparison: Agrylin (Young) vs Agrylin (Elderly); Test type: Superiority or Other; p = 0.013, ANOVA

8. Primary Outcome: Volume of Distribution (Vz/F) of Agrylin
Time Frame: over 1 day
Population: PK population
Measure: Geometric Mean (Standard Deviation); unit: L
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
L | 286 (125) | 195 (137)
Statistical Analysis 1: Comparison: Agrylin (Young) vs Agrylin (Elderly); Test type: Superiority or Other; p = 0.035, ANOVA

9. Primary Outcome: Cmax of Active Metabolite
Description: An active metabolite has therapeutic activity similar to the parent compound and must be considered in therapeutic pharmacokinetics.
Time Frame: over 1 day
Population: PK population
Measure: Geometric Mean (Standard Deviation); unit: ng/ml
Groups:
- Agrylin (Young): Active metabolite of Agrylin (BCH24426) in ages 18-50
- Agrylin (Elderly): Active metabolite of Agrylin (BCH24426) in ages 65 and older
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
ng/ml | 7.26 (3.74) | 4.19 (3.47)
Statistical Analysis 1: Comparison: Agrylin (Young) vs Agrylin (Elderly); Test type: Superiority or Other; p = 0.023, ANOVA

10. Primary Outcome: Tmax of Active Metabolite
Time Frame: over 1 day
Population: PK population
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
hours | 0.92 (0.26) | 1.04 (0.99)
Statistical Analysis 1: Comparison: Agrylin (Young) vs Agrylin (Elderly); Test type: Superiority or Other; p = 0.557, ANOVA

11. Primary Outcome: AUC of Active Metabolite
Time Frame: over 1 day
Population: PK population
Measure: Geometric Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
ng.h/ml | 27.6 (10.9) | 17.4 (14.8)
Statistical Analysis 1: Comparison: Agrylin (Young) vs Agrylin (Elderly); Test type: Superiority or Other; p = 0.027, ANOVA

12. Primary Outcome: T 1/2 of Active Metabolite
Time Frame: over 1 day
Population: PK population
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
hours | 2.7 (0.5) | 3.5 (1.1)
Statistical Analysis 1: Comparison: Agrylin (Young) vs Agrylin (Elderly); Test type: Superiority or Other; p = 0.007, ANOVA

13. Primary Outcome: CL/F of Active Metabolite
Time Frame: over 1 day
Population: PK population
Measure: Geometric Mean (Standard Deviation); unit: L/h
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
L/h | 36 (16) | 57 (27)
Statistical Analysis 1: Comparison: Agrylin (Young) vs Agrylin (Elderly); Test type: Superiority or Other; p = 0.027, ANOVA

14. Primary Outcome: Vz/F of Active Metabolite
Time Frame: over 1 day
Population: PK population
Measure: Geometric Mean (Standard Deviation); unit: L
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
L | 139 (86) | 277 (203)
Statistical Analysis 1: Comparison: Agrylin (Young) vs Agrylin (Elderly); Test type: Superiority or Other; p = 0.011, ANOVA

15. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressures in patients with ET receiving Agrylin
Time Frame: over 1 day
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
mmHg
  Baseline | 122.2 (9.6) | 154.3 (19.6)
  0.5 hours post-dose | 122.7 (12.9) | 145.2 (20.3)
  1.0 hours post-dose | 121.8 (11.7) | 143.7 (21.8)
  1.5 hours post-dose | 122.3 (11.6) | 140.1 (17.7)
  2 hours post-dose | 121.3 (12.3) | 139.9 (19.8)
  4 hours post-dose | 122.2 (13.6) | 133.7 (18.1)
  6 hours post-dose | 120.2 (16.1) | 141.8 (19.5)
  8 hours post-dose | 123.6 (14.5) | 136.3 (24.3)
  12 hours post-dose | 124.7 (13.6) | 159.8 (28.6)

16. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressures in patients with ET receiving Agrylin
Time Frame: over 1 day
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Number analyzed (Participants) | 12 | 12
mmHg
  Baseline | 76.9 (7.5) | 81.4 (10.3)
  0.5 hours post-dose | 74.8 (7.3) | 75.2 (9.9)
  1 hour post-dose | 72.4 (6.6) | 72.6 (7.5)
  1.5 hours post-dose | 72.8 (6.7) | 71.6 (9.5)
  2 hours post-dose | 71.3 (7.9) | 72.8 (7.1)
  4 hours post-dose | 76.2 (6.0) | 73.0 (9.5)
  6 hours post-dose | 73.4 (10.0) | 71.3 (7.6)
  8 hours post-dose | 76.3 (6.2) | 75.0 (11.3)
  12 hours post-dose | 76.3 (9.1) | 84.2 (12.4)

ADVERSE EVENTS:
Arm/Group | Agrylin (Young) | Agrylin (Elderly)
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Agrylin (Young) (N=12) | Agrylin (Elderly) (N=12)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.